CLINICAL TRIAL: NCT05817773
Title: The Design, Development and Effect of Breastfeeding Cradle on Breastfeeding Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehtap Nailoglu, specialist midwife, Ataturk University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: AtaturkU MNailoglu0001
Record Dates: First submitted 2023-02-23; First posted 2023-04-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Women
Keywords: breastfeeding cradle; breastfeeding self-efficacy; postpartum

STUDY DESIGN:
Intervention Model Description: Breastfeeding cradle with remote control system is designed for the mother to breastfeed her baby comfortably. The mother can breastfeed her baby in any position without getting out of bed. Thanks to the remote control, it can give the cradle the desired position. She can safely breastfeed her baby in the cradle with seat belt and safety lock. Breastfeeding cradle with massage, music and light system will provide high comfort for mother and baby.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breastfeeding cradle (Experimental): After the control group was given breastfeeding education and the baby was breastfed, the questionnaire and breastfeeding self-efficacy scale were applied at the 6th hour postoperatively. The experimental group was given breastfeeding education and the baby was placed in a nursing cradle and the baby was breastfed. Then, the questionnaire and breastfeeding self-efficacy scale were applied at the 6th hour postoperatively.
  Interventions: Device: breastfeeding cradle

INTERVENTIONS:
Device: breastfeeding cradle — Mothers with postop mobile cesarean section should be breastfed with a nursing cradle for 30 minutes every 2-3 hours, even if the baby does not cry, until after mobilization (for 6 hours after coming to the service) every time the baby cries.

SUMMARY:
After cesarean section, mothers who are not mobile and cannot take a suitable position to breastfeed their baby, with the designed breastfeeding cradle, the baby approaches the mother's breast and by taking the appropriate position, effective and easy breastfeeding is ensured.

DETAILED DESCRIPTION:
Breastfeeding is considered the most appropriate feeding method because it has many benefits for mother and baby. The benefit of breast milk, which is the most beneficial and unique feeding method for the healthy growth and development of babies biologically, psychologically and emotionally, is indisputable. There is no doubt that breast milk is one of the greatest life savers and that breast milk is a miracle.

Breastfeeding within the first half hour after birth is one of the Baby-Friendly Hospital criteria, a program of the World Health Organization (WHO) and the United Nations International Children's Emergency Fund (UNICEF). The baby's active period after birth is the first half hour. In this process, breastfeeding affects the success of breastfeeding and the duration of breastfeeding positively. Failure to start breastfeeding in the early postpartum period and the lack of a successful breastfeeding process can have important consequences for the health of the mother and baby in the short and long term. WHO states that breastfeeding in the first half-hour period after birth reduces the risk of death and disease in infants, and then increases breastfeeding rates. International and national organizations have stated that breastfeeding of mothers in the first half-hour period after birth increases the probability of survival of babies, skin-to-skin contact is achieved earlier, increases milk production, including colostrum, and increases uterine involution.

There has been a significant increase in cesarean section rates in our country as well as in the world in recent years. According to Turkey Demographic Health Survey (TNSA) 2018 data, cesarean deliveries account for 52% of all deliveries in Turkey. Mothers with cesarean section experience more problems with breastfeeding compared to mothers who gave birth normally. Some of the most important problems with breastfeeding after cesarean section are that mothers have difficulty breastfeeding without the help of someone due to the limitation of movement after cesarean section. Another problem experienced in the early postpartum period after cesarean section is that mothers may not want to breastfeed their babies because of the concern that the baby will experience pain after the baby's contact instead of the cesarean section incision while breastfeeding. Expecting the mother to be mobile for the first breastfeeding negatively affects breastfeeding self-efficacy. The need for support is higher in cesarean deliveries than in normal births. For this, there must be sufficient midwives who can be sufficient here. It is thought that the most important factor in the failure of breastfeeding after cesarean section is the wrong breastfeeding position. In order for breastfeeding to be easier and more comfortable, the tools produced to support breastfeeding should be useful, easy and effective in breastfeeding. Tools used in breastfeeding self-efficacy; breastfeeding support system, breastfeeding pillow, breastfeeding apron and breastfeeding chair.

ELIGIBILITY:
Inclusion Criteria:

18- 35 years old, Primipar, At least primary school graduate, No high-risk pregnancy Absence of any complications in the birth and postpartum period in the newborn and himself.

Exclusion Criteria:

Those who have any contraindication for breastfeeding Having a baby under 3000 g, Mothers whose baby was not with them due to any health reasons were not included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primipar puerperant women
Enrollment: 141 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The effect of breastfeeding cradle on breastfeeding self-efficacy | seven months
  breastfeeding cradle is effective on breastfeeding self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Serap EJDER APAY, prof, Principal Investigator — ataturk university midwifery department
Locations (1):
- Atatürk Unıversıty, Erzurum, Erzurum/Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not a plan for use of individual participant data (IPD) by other researchers.